CLINICAL TRIAL: NCT00024128
Title: Delayed Donor Leukocyte Infusions in Patients Receiving Allogeneic PBSC Following Conditioning With Non-myeloablative Regimen for AIDS-Related Lymphoma (NHL and HD)
Brief Title: Peripheral Stem Cell Transplantation Followed By Infusion of White Blood Cells in Treating Patients With AIDS-Related Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn prior to initiation.
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-028; CDR0000068894 (Other: NCI)
Record Dates: First submitted 2001-09-13; First posted 2003-10-21 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma; HIV-associated Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Antilymphocyte Serum; Cyclophosphamide; Cyclosporine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: therapeutic allogeneic lymphocytes
Drug: cyclophosphamide
Drug: cyclosporine
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Donor peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy. Sometimes the transplanted cells are rejected by the body's normal tissues. Treatment with donor white blood cells may prevent this from happening.

PURPOSE: Phase II trial to study the effectiveness of donor peripheral stem cell transplantation followed by infusions of donor white blood cells in treating patients who have AIDS-related lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with AIDS-related lymphoma treated with allogeneic peripheral blood stem cell (PBSC) transplantation followed by delayed donor leukocyte infusion.
* Determine the complication rate of these patients treated with PBSC transplantation.
* Determine the immune dysfunction and recovery of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive cyclophosphamide IV over 60 minutes on days -5 to -3. Patients who have not received prior mediastinal radiotherapy receive thymic radiotherapy on day -1. Allogeneic peripheral blood stem cells are infused on day 0. Patients also receive anti-thymocyte globulin IV over 10-12 hours on days -1, 1, 3, and 5 and cyclosporine IV beginning on day -1, switching to oral when possible, and tapering until day 35.

In the absence of active acute graft-versus-host disease (GVHD), and at least 2 weeks after completion of cyclosporine, patients receive an infusion of donor leukocytes on or before day 49. Patients may receive a second donor leukocyte infusion if there is evidence of persistent malignancy and no GVHD.

Patients are followed through day 100, on days 120, 180, 270, and 365, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 12-35 patients will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Hodgkin's disease or non-Hodgkin's lymphoma

  * Failed to achieve a complete remission with initial therapy OR
  * Relapsed after initial therapy
* HIV-1 seropositive by Western Blot
* Measurable or evaluable (e.g., pleural fluid involvement) disease
* No leptomeningeal or parenchymal CNS involvement or active CNS leukemia
* HLA-A, B, or DR antigen matched or 1 antigen mismatched related donor available
* CD4 cell count greater than 100/mm3 (initial 12 patients) OR greater than 50/mm3 (subsequent patients)*
* HIV RNA less than 110,000 copies/mL* NOTE: *Unless not receiving optimal anti-retroviral therapy as defined by current clinical standards

PATIENT CHARACTERISTICS:

Age:

* Physiologic 65 and under

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Estimated disease-free survival less than 1 year

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2 mg/dL
* Alkaline phosphatase no greater than 3 times upper limit of normal (ULN)*
* SGOT or SGPT no greater than 3 times ULN*
* Hepatitis B surface antigen negative NOTE: *Unless receiving indinavir

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No angina pectoris
* No uncontrolled hypertension
* LVEF at least 45% by radionuclide ventriculography

Pulmonary:

* No severe chronic obstructive lung disease
* No symptomatic restrictive lung disease
* DLCO greater than 50% predicted

Other:

* No active uncontrolled infection
* No history of cytomegalovirus retinitis or pneumonitis, even if treated
* No other disease that would limit life expectancy
* No symptomatic leukoencephalopathy
* No neuropsychiatric abnormalities that would preclude transplantation
* Human T-cell lymphotrophic virus (HTLV-1) antibody negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 1 week since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent chronic suppressive therapy

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-08; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T. Scadden, MD, Study Chair — Massachusetts General Hospital